CLINICAL TRIAL: NCT00688870
Title: A PHASE 3, RANDOMIZED, ACTIVE-CONTROLLED, DOUBLE-BLIND TRIAL EVALUATING THE SAFETY, TOLERABILITY AND IMMUNOGENICITY OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS GIVEN WITH ROUTINE PEDIATRIC VACCINATION IN TAIWAN
Brief Title: Study Evaluating A 13-Valent Pneumococcal Conjugate Vaccine Administered to Infants in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-3004; B1851005 (Other: Alias Study Number); 2008-004766-40 (EudraCT Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2011-05-12 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Vaccines; Pneumococcal Conjugate Vaccine
Keywords: Prevention against pneumococcal disease
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 13vPnC
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)
- 2 (Active Comparator): 7vPnC
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine (7vPnC)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 13vPnC is given via intramuscular injection at approximately 2, 4, 6, and 15 months of age.
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine (7vPnC) — 7vPnC is given via intramuscular injection at approximately 2, 4, 6, and 15 months of age.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate vaccine (13vPnC), relative to a 7-valent pneumococcal conjugate vaccine (7vPnC) when given concomitantly with routine vaccines in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old infants (42 to 98 days)
* Available for the entire study period (14 months)

Exclusion Criteria:

* Previous vaccination with pneumococcal, diphtheria, tetanus, pertussis, polio, or Hib vaccines
* A previous anaphylactic reaction to any vaccine or vaccine-related component.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-06-05 (Actual); Primary Completion 2010-01-13 (Actual); Study Completion 2010-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linko, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Huang LM, Lin TY, Juergens C. Immunogenicity and safety of a 13-valent pneumococcal conjugate vaccine given with routine pediatric vaccines in Taiwan. Vaccine. 2012 Mar 9;30(12):2054-9. doi: 10.1016/j.vaccine.2011.12.054. Epub 2011 Dec 22. PMID 22198517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Taiwan from June 2008 to Nov 2009
Pre-assignment Details: A total of 169 subjects were screened, 168 subjects were randomly assigned in a 1:1 ratio to either the 13vPnC group (n=84) or the 7vPnC group (n=84).
Groups:
- 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly, at 2, 4 and 6 months of age (infant series) and 15 months of age (toddler dose). At 2 and 4 months of age during the infant series, 13vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, and acellular pertussis (DTaP); inactivated poliovirus (IPV); and H influenzae type b (Hib). At 6 months of age during the infant series, 13vPnC was co-administered with DTaP-IPV-Hib and hepatitis B virus (HBV) vaccine.
- 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 2, 4 and 6 months of age (infant series) and 15 months of age (toddler dose). At 2 and 4 months of age during the infant series, 7vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, and acellular pertussis (DTaP); inactivated poliovirus (IPV); and H influenzae type b (Hib). At 6 months of age during the infant series, 7vPnC was co-administered with DTaP-IPV-Hib and hepatitis B virus (HBV) vaccine.
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 84 | 84
Vaccinated Dose 1 | 83 | 84
Vaccinated Dose 2 | 80 | 84
Vaccinated Dose 3 | 80 | 84
Completed | 80 | 84
Not Completed | 4 | 0
Not completed — Parent or legal guardian request | 4 | 0
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 80 | 84
Completed | 80 | 84
Not Completed | 0 | 0
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 80 | 84
Completed | 80 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC: Participants received 1 single 0.5 mL dose of 13vPnC, administered intramuscularly, at 2, 4 and 6 months of age (infant series) and 15 months of age (toddler dose). At 2 and 4 months of age during the infant series, 13vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, and acellular pertussis (DTaP); inactivated poliovirus (IPV); and H influenzae type b (Hib). At 6 months of age during the infant series, 13vPnC was co-administered with DTaP-IPV-Hib and hepatitis B virus (HBV) vaccine.
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.2 (0.3) | 2.3 (0.3) | 2.2 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 44 | 37 | 81
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan, Province Of China | 84 | 84 | 168

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Predefined Antibody Level of Greater Than or Equal to 0.35 Micrograms (mcg)/mL, 1 Month After the Infant Series.
Description: Percentage of participants achieving a predefined antibody level of greater than or equal to 0.35 mcg/mL along with the corresponding exact 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all 3 doses, blood drawn within specified timeframes, had at least 1 valid and determinate assay result for the proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 83
percentage of participants
  Common Serotypes - Serotype 4 | 98.8 [93.2 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 6B | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 9V | 98.8 [93.2 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 14 | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 18C | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 19F | 98.8 [93.2 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 23F | 95.0 [87.7 to 98.6] | 100.0 [95.7 to 100.0]
  Additional Serotypes - Serotype 1 | 98.8 [93.2 to 100.0] | 2.4 [0.3 to 8.4]
  Additional Serotypes - Serotype 3 | 97.5 [91.3 to 99.7] | 2.4 [0.3 to 8.4]
  Additional Serotypes - Serotype 5 | 98.8 [93.2 to 100.0] | 61.5 [49.8 to 72.3]
  Additional Serotypes - Serotype 6A | 100.0 [95.5 to 100.0] | 77.1 [66.6 to 85.6]
  Additional Serotypes - Serotype 7F | 100.0 [95.5 to 100.0] | 2.4 [0.3 to 8.4]
  Additional Serotypes - Serotype 19A | 100.0 [95.5 to 100.0] | 100.0 [95.6 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — Exact, unconditional, 2-sided 95% CI for the difference in proportions were computed using the noninferiority procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Chan and Zhang; Difference = -1.2, 95% CI 2-sided [-6.8 to 3.3]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.3]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -1.2, 95% CI 2-sided [-6.8 to 3.3]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.3]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.3]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -1.2, 95% CI 2-sided [-6.8 to 3.3]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -5.0, 95% CI 2-sided [-12.3 to -0.3]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 96.3, 95% CI 2-sided [89.4 to 99.2]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 95.1, 95% CI 2-sided [87.7 to 98.6]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 37.2, 95% CI 2-sided [26.2 to 48.9]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 22.9, 95% CI 2-sided [14.4 to 33.4]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 97.6, 95% CI 2-sided [91.6 to 99.7]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.5]

2. Secondary Outcome: Percentage of Participants Achieving a Predefined Antibody Level of Greater Than or Equal to 0.35 mcg/mL, 1 Month After the Toddler Dose
Description: Percentage of participants achieving a predefined antibody level of greater than or equal to 0.35 mcg/mL along with the corresponding exact 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 month after toddler dose (16 months of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all 4 doses, blood drawn within specified timeframes, had at least 1 valid and determinate assay result for the proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 79 | 84
percentage of participants
  Common Serotypes - Serotype 4 | 98.7 [93.1 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 6B | 100.0 [95.4 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 9V | 98.7 [93.1 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 14 | 100.0 [95.4 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 18C | 100.0 [95.4 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 19F | 98.7 [93.1 to 100.0] | 100.0 [95.7 to 100.0]
  Common Serotypes - Serotype 23F | 100.0 [95.4 to 100.0] | 100.0 [95.7 to 100.0]
  Additional Serotypes - Serotype 1 | 100.0 [95.4 to 100.0] | 5.0 [1.4 to 12.3]
  Additional Serotypes - Serotype 3 | 96.2 [89.3 to 99.2] | 13.8 [7.1 to 23.3]
  Additional Serotypes - Serotype 5 | 100.0 [95.4 to 100.0] | 90.4 [81.9 to 95.7]
  Additional Serotypes - Serotype 6A | 100.0 [95.4 to 100.0] | 100.0 [95.7 to 100.0]
  Additional Serotypes - Serotype 7F | 100.0 [95.4 to 100.0] | 6.3 [2.1 to 14.0]
  Additional Serotypes - Serotype 19A | 100.0 [95.4 to 100.0] | 98.8 [93.5 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -1.3, 95% CI 2-sided [-6.9 to 3.1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -1.3, 95% CI 2-sided [-6.9 to 3.1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = -1.3, 95% CI 2-sided [-6.9 to 3.1]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 95.0, 95% CI 2-sided [87.7 to 98.6]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 82.5, 95% CI 2-sided [72.0 to 90.1]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 9.6, 95% CI 2-sided [3.8 to 18.1]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 0.0, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 93.8, 95% CI 2-sided [86.0 to 97.9]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Chan and Zhang; Difference = 1.2, 95% CI 2-sided [-3.4 to 6.5]

3. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody, 1 Month After the Infant Series
Description: Antibody GMC as measured in mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: GMC mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 83
GMC mcg/mL
  Common serotypes - serotype 4 | 2.89 [2.45 to 3.42] | 4.64 [4.00 to 5.37]
  Common serotypes - serotype 6B | 4.37 [3.58 to 5.33] | 4.82 [4.09 to 5.67]
  Common serotypes - serotype 9V | 1.97 [1.70 to 2.27] | 2.92 [2.55 to 3.34]
  Common serotypes - serotype 14 | 9.76 [8.34 to 11.43] | 11.59 [9.79 to 13.71]
  Common serotypes - serotype 18C | 2.39 [2.04 to 2.82] | 3.07 [2.64 to 3.56]
  Common serotypes - serotype 19F | 3.60 [3.00 to 4.32] | 4.77 [4.17 to 5.47]
  Common serotypes - serotype 23F | 1.93 [1.56 to 2.37] | 3.25 [2.78 to 3.80]
  Additional serotypes - serotype 1 | 4.14 [3.45 to 4.96] | 0.02 [0.02 to 0.02]
  Additional serotypes - serotype 3 | 1.20 [1.00 to 1.45] | 0.05 [0.04 to 0.06]
  Additional serotypes - serotype 5 | 2.47 [2.09 to 2.92] | 0.43 [0.35 to 0.53]
  Additional serotypes - serotype 6A | 4.57 [3.92 to 5.34] | 0.79 [0.63 to 0.99]
  Additional serotypes - serotype 7F | 3.67 [3.14 to 4.29] | 0.04 [0.03 to 0.05]
  Additional serotypes - serotype 19A | 3.69 [3.20 to 4.24] | 2.46 [2.13 to 2.84]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 4; Test type: Superiority or Other; ratio of GMCs = 0.62, 95% CI 2-sided [0.50 to 0.78] — Confidence intervals for the ratio are back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC-7vPnC reference)
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 6B; Test type: Superiority or Other; ratio of GMCs = 0.91, 95% CI 2-sided [0.70 to 1.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 9V; Test type: Superiority or Other; ratio of GMCs = 0.67, 95% CI 2-sided [0.55 to 0.82] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 14; Test type: Superiority or Other; ratio of GMCs = 0.84, 95% CI 2-sided [0.67 to 1.06] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 18C; Test type: Superiority or Other; ratio of GMCs = 0.78, 95% CI 2-sided [0.63 to 0.97] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 19F; Test type: Superiority or Other; ratio of GMCs = 0.75, 95% CI 2-sided [0.60 to 0.94] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 23F; Test type: Superiority or Other; ratio of GMCs = 0.59, 95% CI 2-sided [0.46 to 0.77] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 1; Test type: Superiority or Other; ratio of GMCs = 202.58, 95% CI 2-sided [157.04 to 261.32] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 3; Test type: Superiority or Other; ratio of GMCs = 24.11, 95% CI 2-sided [18.46 to 31.49] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 5; Test type: Superiority or Other; ratio of GMCs = 5.69, 95% CI 2-sided [4.37 to 7.41] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 6A; Test type: Superiority or Other; ratio of GMCs = 5.82, 95% CI 2-sided [4.42 to 7.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 7F; Test type: Superiority or Other; ratio of GMCs = 96.10, 95% CI 2-sided [75.60 to 122.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 19A; Test type: Superiority or Other; ratio of GMCs = 1.50, 95% CI 2-sided [1.23 to 1.83] — [estimate comment as in outcome 3, analysis 1]

4. Other Pre Specified Outcome: GMC for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody, 1 Month After the Toddler Dose
Description: as for outcome 3
Time Frame: 1 month after the toddler dose (16 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: GMC mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 79 | 84
GMC mcg/mL
  Common serotypes - serotype 4 | 4.06 [3.34 to 4.93] | 6.34 [5.26 to 7.65]
  Common serotypes - serotype 6B | 13.62 [11.08 to 16.73] | 13.28 [10.87 to 16.21]
  Common serotypes - serotype 9V | 3.18 [2.66 to 3.80] | 3.88 [3.27 to 4.60]
  Common serotypes - serotype 14 | 8.17 [6.53 to 10.22] | 12.04 [9.90 to 14.63]
  Common serotypes - serotype 18C | 3.67 [3.00 to 4.49] | 4.87 [4.01 to 5.90]
  Common serotypes - serotype 19F | 8.07 [6.58 to 9.90] | 7.41 [6.16 to 8.92]
  Common serotypes - serotype 23F | 5.51 [4.46 to 6.81] | 7.97 [6.55 to 9.68]
  Additional serotypes - serotype 1 | 7.62 [6.30 to 9.21] | 0.03 [0.02 to 0.03]
  Additional serotypes - serotype 3 | 1.29 [1.09 to 1.53] | 0.12 [0.09 to 0.16]
  Additional serotypes - serotype 5 | 4.57 [3.87 to 5.39] | 0.95 [0.80 to 1.13]
  Additional serotypes - serotype 6A | 11.55 [9.66 to 13.81] | 3.79 [3.01 to 4.76]
  Additional serotypes - serotype 7F | 5.91 [4.95 to 7.06] | 0.06 [0.04 to 0.07]
  Additional serotypes - serotype 19A | 8.82 [7.45 to 10.43] | 1.98 [1.69 to 2.32]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 4; Test type: Superiority or Other; ratio of GMC = 0.64, 95% CI 2-sided [0.49 to 0.84] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 6B; Test type: Superiority or Other; ratio of GMCs = 1.03, 95% CI 2-sided [0.77 to 1.36] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 9V; Test type: Superiority or Other; ratio of GMCs = 0.82, 95% CI 2-sided [0.64 to 1.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 14; Test type: Superiority or Other; ratio of GMCs = 0.68, 95% CI 2-sided [0.51 to 0.91] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 18C; Test type: Superiority or Other; ratio of GMCs = 0.75, 95% CI 2-sided [0.57 to 0.99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 19F; Test type: Superiority or Other; ratio of GMCs = 1.09, 95% CI 2-sided [0.83 to 1.43] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Common serotypes - serotype 23F; Test type: Superiority or Other; ratio of GMCs = 0.69, 95% CI 2-sided [0.52 to 0.92] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 1; Test type: Superiority or Other; ratio of GMCs = 303.73, 95% CI 2-sided [213.63 to 431.83] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 3; Test type: Superiority or Other; ratio of GMCs = 10.65, 95% CI 2-sided [7.77 to 14.62] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 5; Test type: Superiority or Other; ratio of GMCs = 4.79, 95% CI 2-sided [3.78 to 6.08] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 6A; Test type: Superiority or Other; ratio of GMCs = 3.05, 95% CI 2-sided [2.28 to 4.08] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 7F; Test type: Superiority or Other; ratio of GMCs = 105.00, 95% CI 2-sided [75.60 to 145.84] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Additional serotypes - serotype 19A; Test type: Superiority or Other; ratio of GMCs = 4.45, 95% CI 2-sided [3.54 to 5.60] — [estimate comment as in outcome 3, analysis 1]

5. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 1 (2 Months of Age).
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling and redness present); Mild (0.5 to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after Dose 1 of the infant series (2 Months of Age)
Population: Safety population: all participants who received dose 1 of the infant series vaccination (2 months of age). number analyzed= number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 83 | 84
percentage of participants
  Tenderness - Any | 31.3 | 34.2
  Tenderness - Significant | 5.3 | 9.3
  Swelling - Any | 25.6 | 11.8
  Swelling - Mild | 24.4 | 11.8
  Swelling - Moderate: number analyzed (Participants) | 74 | 74
  Swelling - Moderate | 1.4 | 0.0
  Swelling - Severe: number analyzed (Participants) | 74 | 74
  Swelling - Severe | 0.0 | 0.0
  Redness - Any | 29.9 | 28.9
  Redness - Mild | 26.0 | 26.3
  Redness - Moderate: number analyzed (Participants) | 74 | 74
  Redness - Moderate | 8.1 | 2.7
  Redness - Severe: number analyzed (Participants) | 74 | 74
  Redness - Severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Tenderness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.735, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Tenderness - Significant, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.533, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Swelling - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.039, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Swelling - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.059, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Swelling - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Redness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Redness - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For Redness - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.275, Fisher Exact

6. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 5
Time Frame: Within 4 Days after Dose 2 of the infant series (4 months of age)
Population: Safety population: all participants who received the first 2 doses of the infant series vaccination (4 months of age). n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Tenderness - Any | 23.6 | 22.4
  Tenderness - Significant: number analyzed (Participants) | 69 | 71
  Tenderness - Significant | 2.9 | 1.4
  Swelling - Any: number analyzed (Participants) | 70 | 72
  Swelling - Any | 12.9 | 15.3
  Swelling - Mild: number analyzed (Participants) | 70 | 72
  Swelling - Mild | 12.9 | 15.3
  Swelling - Moderate: number analyzed (Participants) | 69 | 71
  Swelling - Moderate | 0.0 | 0.0
  Swelling - Severe: number analyzed (Participants) | 69 | 71
  Swelling - Severe | 0.0 | 0.0
  Redness - Any: number analyzed (Participants) | 70 | 74
  Redness - Any | 17.1 | 20.3
  Redness - Mild: number analyzed (Participants) | 70 | 74
  Redness - Mild | 17.1 | 17.6
  Redness - Moderate: number analyzed (Participants) | 69 | 71
  Redness - Moderate | 0.0 | 2.8
  Redness - Severe: number analyzed (Participants) | 69 | 71
  Redness - Severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Tenderness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Tenderness - Significant, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.617, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Swelling - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.810, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Swelling - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.810, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Redness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.674, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Redness - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Redness - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.497, Fisher Exact

7. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 5
Time Frame: Within 4 days after Dose 3 of the infant series (6 months of age)
Population: Safety population: all participants who received all 3 doses of the infant series vaccination (6 months of age). n=number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Tenderness - Any: number analyzed (Participants) | 67 | 67
  Tenderness - Any | 19.4 | 17.9
  Tenderness - Significant: number analyzed (Participants) | 65 | 65
  Tenderness - Significant | 0.0 | 1.5
  Swelling - Any: number analyzed (Participants) | 65 | 65
  Swelling - Any | 16.9 | 4.6
  Swelling - Mild: number analyzed (Participants) | 65 | 65
  Swelling - Mild | 15.4 | 4.6
  Swelling - Moderate: number analyzed (Participants) | 65 | 64
  Swelling - Moderate | 3.1 | 0.0
  Swelling - Severe: number analyzed (Participants) | 65 | 64
  Swelling - Severe | 0.0 | 0.0
  Redness - Any: number analyzed (Participants) | 67 | 65
  Redness - Any | 20.9 | 13.8
  Redness - Mild: number analyzed (Participants) | 66 | 65
  Redness - Mild | 18.2 | 13.8
  Redness - Moderate: number analyzed (Participants) | 66 | 64
  Redness - Moderate | 4.5 | 0.0
  Redness - Severe: number analyzed (Participants) | 65 | 64
  Redness - Severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Tenderness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Tenderness - Significant, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Swelling - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.044, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Swelling - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.076, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Swelling - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.496, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Redness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.361, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Redness - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.635, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For Redness - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.244, Fisher Exact

8. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Toddler Dose (15 Months of Age).
Description: as for outcome 5
Time Frame: Within 4 days after the toddler dose (15 months of age)
Population: Safety population: all participants who received the toddler dose (15 months of age). n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Tenderness - Any: number analyzed (Participants) | 64 | 75
  Tenderness - Any | 10.9 | 22.7
  Tenderness - Significant: number analyzed (Participants) | 63 | 69
  Tenderness - Significant | 0.0 | 0.0
  Swelling - Any: number analyzed (Participants) | 63 | 70
  Swelling - Any | 7.9 | 5.7
  Swelling - Mild: number analyzed (Participants) | 63 | 70
  Swelling - Mild | 6.3 | 5.7
  Swelling - Moderate: number analyzed (Participants) | 63 | 69
  Swelling - Moderate | 1.6 | 0.0
  Swelling - Severe: number analyzed (Participants) | 63 | 69
  Swelling - Severe | 0.0 | 0.0
  Redness - Any: number analyzed (Participants) | 65 | 70
  Redness - Any | 15.4 | 12.9
  Redness - Mild: number analyzed (Participants) | 65 | 70
  Redness - Mild | 13.8 | 12.9
  Redness - Moderate: number analyzed (Participants) | 63 | 69
  Redness - Moderate | 1.6 | 0.0
  Redness - Severe: number analyzed (Participants) | 63 | 69
  Redness - Severe | 0.0 | 0.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Tenderness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.076, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Swelling - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.735, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Swelling - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Swelling - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.477, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Redness - Any, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.805, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Redness - Mild, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Redness - Moderate, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.477, Fisher Exact

9. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 1 (2 Months of Age)
Description: Systemic events (any fever >=38 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after Dose 1 of the infant series (2 months of age)
Population: Safety population: all participants who received dose 1 of the infant series vaccination (2 months of age). (n)= number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 83 | 84
percentage of participants
  Fever >=38 but <=39 degrees C | 55.0 | 50.0
  Fever >39 but <=40 degrees C: number analyzed (Participants) | 74 | 74
  Fever >39 but <=40 degrees C | 1.4 | 1.4
  Fever >40 degrees C: number analyzed (Participants) | 74 | 74
  Fever >40 degrees C | 0.0 | 0.0
  Decreased appetite | 50.0 | 55.6
  Irritability | 65.0 | 70.0
  Increased sleep | 53.2 | 50.6
  Decreased sleep | 44.3 | 41.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Fever >=38 but <=39 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.633, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Fever >39 but <=40 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Decreased appetite, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.527, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Irritability, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.613, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Increased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.753, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Decreased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.748, Fisher Exact

10. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 2 (4 Months of Age)
Description: Systemic events (any fever >=38 degrees C, decreased appetite, irritability, increased sleep, decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after Dose 2 of the infant series (4 months of age)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Fever >=38 but <=39 degrees C | 52.1 | 43.4
  Fever >39 but <=40 degrees C: number analyzed (Participants) | 69 | 72
  Fever >39 but <=40 degrees C | 2.9 | 2.8
  Fever >40 degrees C: number analyzed (Participants) | 69 | 71
  Fever >40 degrees C | 0.0 | 0.0
  Decreased appetite | 50.7 | 56.1
  Irritability | 56.0 | 57.5
  Increased sleep | 41.1 | 43.4
  Decreased sleep: number analyzed (Participants) | 71 | 77
  Decreased sleep | 42.3 | 32.5
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Fever >=38 but <=39 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.327, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Fever >39 but <=40 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Decreased appetite, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.522, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Irritability, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.872, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Increased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.868, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Decreased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.237, Fisher Exact

11. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 10
Time Frame: Within 4 days after dose 3 of the infant series (6 months of age)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Fever >=38 but <=39 degrees C: number analyzed (Participants) | 66 | 66
  Fever >=38 but <=39 degrees C | 31.8 | 22.7
  Fever >39 but <=40 degrees C: number analyzed (Participants) | 65 | 66
  Fever >39 but <=40 degrees C | 4.6 | 9.1
  Fever >40 degrees C: number analyzed (Participants) | 65 | 64
  Fever >40 degrees C | 0.0 | 1.6
  Decreased appetite: number analyzed (Participants) | 69 | 75
  Decreased appetite | 43.5 | 52.0
  Irritability: number analyzed (Participants) | 68 | 71
  Irritability | 42.6 | 47.9
  Increased sleep: number analyzed (Participants) | 66 | 70
  Increased sleep | 40.9 | 37.1
  Decreased sleep: number analyzed (Participants) | 68 | 69
  Decreased sleep | 30.9 | 33.3
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Fever >=38 but <=39 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.329, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Fever >39 but <=40 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.492, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Fever >40 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.496, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Decreased appetite, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.322, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Irritability, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.610, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Increased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.726, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Decreased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.855, Fisher Exact

12. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Toddler Dose (15 Months of Age).
Description: as for outcome 10
Time Frame: Within 4 days after the toddler dose (15 months of age)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 80 | 84
percentage of participants
  Fever >=38 but <=39 degrees C: number analyzed (Participants) | 65 | 70
  Fever >=38 but <=39 degrees C | 29.2 | 21.4
  Fever >39 but <=40 degrees C: number analyzed (Participants) | 63 | 69
  Fever >39 but <=40 degrees C | 3.2 | 4.3
  Fever >40 degrees C: number analyzed (Participants) | 63 | 69
  Fever >40 degrees C | 0.0 | 0.0
  Decreased appetite: number analyzed (Participants) | 65 | 75
  Decreased appetite | 27.7 | 30.7
  Irritability: number analyzed (Participants) | 65 | 74
  Irritability | 27.7 | 27.0
  Increased sleep: number analyzed (Participants) | 66 | 72
  Increased sleep | 16.7 | 16.7
  Decreased sleep: number analyzed (Participants) | 64 | 74
  Decreased sleep | 17.2 | 23.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Fever >=38 but <=39 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.326, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Fever >39 but <=40 degrees C, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Decreased appetite, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.714, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Irritability, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Increased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Decreased sleep, Fisher exact test was used to calculate p-value; Test type: Superiority or Other; p = 0.525, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 1 month after last study vaccination (16 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1=2 months of age; Dose 2=4 months of age; Dose 3=6 months of age; Toddler Dose=15 months of age.
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event
Groups:
- Infant Series 13vPnC; After the Infant Series 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly, at 2, 4 and 6 months of age (infant series). At 2 and 4 months of age during the infant series, 13vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, and acellular pertussis (DTaP); inactivated poliovirus (IPV); and H influenzae type b (Hib). At 6 months of age during the infant series, 13vPnC was co-administered with DTaP-IPV-Hib and hepatitis B virus (HBV) vaccine.
- Infant Series 7vPnC; After the Infant Series 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 2, 4 and 6 months of age (infant series). At 2 and 4 months of age during the infant series, 7vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, and acellular pertussis (DTaP); inactivated poliovirus (IPV); and H influenzae type b (Hib). At 6 months of age during the infant series, 7vPnC was co-administered with DTaP-IPV-Hib and hepatitis B virus (HBV) vaccine.
- Toddler Dose 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly, at 15 months of age (toddler dose).
- Toddler Dose 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 15 months of age (toddler dose).
Arm/Group | Infant Series 13vPnC | Infant Series 7vPnC | After the Infant Series 13vPnC | After the Infant Series 7vPnC | Toddler Dose 13vPnC | Toddler Dose 7vPnC
Serious Adverse Events (participants affected / at risk) | 4/83 | 4/84 | 12/83 | 9/84 | 0/80 | 3/84
Other Adverse Events (participants affected / at risk) | 81/83 | 77/84 | 11/83 | 16/84 | 39/80 | 47/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=83) | Infant Series 7vPnC (N=84) | After the Infant Series 13vPnC (N=83) | After the Infant Series 7vPnC (N=84) | Toddler Dose 13vPnC (N=80) | Toddler Dose 7vPnC (N=84)
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Roseola (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Testicular retraction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (N=83) | Infant Series 7vPnC (N=84) | After the Infant Series 13vPnC (N=83) | After the Infant Series 7vPnC (N=84) | Toddler Dose 13vPnC (N=80) | Toddler Dose 7vPnC (N=84)
Tenderness (any) (Skin and subcutaneous tissue disorders) | 25/80 | 26/76 | 0/0 | 0/0 | 7/64 | 17/75 — Infant Series Dose 1 and Toddler Dose; Tenderness (any) = present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 17/72 | 17/76 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; tenderness (any) = present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 13/67 | 12/67 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; tenderness (any) = present at site of vaccination.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 4/75 | 7/75 | 0/0 | 0/0 | 0/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant) = present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 2/69 | 1/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant) = present and interfered with limb movement.
Tenderness (signficant) (Skin and subcutaneous tissue disorders) | 0/65 | 1/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant) = present and interfered with limb movement.
Swelling (any) (Skin and subcutaneous tissue disorders) | 20/78 | 9/76 | 0/0 | 0/0 | 5/63 | 4/70 — Infant Series Dose 1 and Toddler Dose; Swelling (any) = present at site of vaccination.
Swelling (any) (Skin and subcutaneous tissue disorders) | 9/70 | 11/72 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (any) = present at site of vaccination.
Swelling (any) (Skin and subcutaneous tissue disorders) | 11/65 | 3/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (any) = present at site of vaccination.
Swelling (mild) (Skin and subcutaneous tissue disorders) | 19/78 | 9/76 | 0/0 | 0/0 | 4/63 | 4/70 — Infant Series Dose 1 and Toddler Dose; Swelling (mild) = 0.5 to 2.0 cm
Swelling (mild) (Skin and subcutaneous tissue disorders) | 9/70 | 11/72 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (mild) = 0.5 to 2.0 cm
Swelling (mild) (Skin and subcutaneous tissue disorders) | 10/65 | 3/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (mild) = 0.5 to 2.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 1/74 | 0/74 | 0/0 | 0/0 | 1/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Swelling (moderate) = 2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 0/69 | 0/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (moderate) = 2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 2/65 | 0/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (moderate) = 2.5 to 7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/74 | 0/74 | 0/0 | 0/0 | 0/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Swelling (severe) = >7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/69 | 0/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (severe) = >7.0 cm
Redness (any) (Skin and subcutaneous tissue disorders) | 23/77 | 22/76 | 0/0 | 0/0 | 10/65 | 9/70 — Infant Series Dose 1 and Toddler Dose; Redness (any) = present at site of vaccination.
Redness (any) (Skin and subcutaneous tissue disorders) | 12/70 | 15/74 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (any) = present at site of vaccination.
Redness (any) (Skin and subcutaneous tissue disorders) | 14/67 | 9/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (any) = present at site of vaccination.
Redness (mild) (Skin and subcutaneous tissue disorders) | 20/77 | 20/76 | 0/0 | 0/0 | 9/65 | 9/70 — Infant Series Dose 1 and Toddler Dose; Redness (mild) = 0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 12/70 | 13/74 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (mild) = 0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 12/66 | 9/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (mild) = 0.5 to 2.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 6/74 | 2/74 | 0/0 | 0/0 | 1/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Redness (moderate) = 2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 0/69 | 2/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (moderate) = 2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 3/66 | 0/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (moderate) = 2.5 to 7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/74 | 0/74 | 0/0 | 0/0 | 0/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Redness (severe) = >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/69 | 0/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (severe) = >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/65 | 0/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (severe) = >7.0 cm
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 44/80 | 39/78 | 0/0 | 0/0 | 19/65 | 15/70 — Infant Series Dose 1 and Toddler Dose; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 38/73 | 33/76 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 21/66 | 15/66 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 1/74 | 1/74 | 0/0 | 0/0 | 2/63 | 3/69 — Infant Series Dose 1 and Toddler Dose; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 2/69 | 2/72 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 3/65 | 6/66 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 40 degrees C (General disorders) | 0/74 | 0/74 | 0/0 | 0/0 | 0/63 | 0/69 — Infant Series Dose 1 and Toddler Dose; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/69 | 0/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/65 | 1/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 40 degrees C
Decreased appetite (General disorders) | 39/78 | 45/81 | 0/0 | 0/0 | 18/65 | 23/75 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 37/73 | 46/82 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 30/69 | 39/75 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 52/80 | 56/80 | 0/0 | 0/0 | 18/65 | 20/74 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 42/75 | 46/80 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 29/68 | 34/71 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 41/77 | 41/81 | 0/0 | 0/0 | 11/66 | 12/72 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 30/73 | 33/76 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 27/66 | 26/70 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 35/79 | 32/78 | 0/0 | 0/0 | 11/64 | 17/74 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 30/71 | 25/77 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 21/68 | 23/69 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/65 | 0/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (severe) = >7.0 cm
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 2 | 0 | 0 | 2 | 2
Milk allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 31 | 53 | 0 | 0 | 9 | 8
Bronchiolitis (Infections and infestations) | 4 | 4 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 7 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 5 | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 3 | 0 | 0 | 1 | 0
Roseola (Infections and infestations) | 3 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 10 | 11 | 5 | 11 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 6 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 5 | 3 | 7 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 3 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Geometric Mean Concentration Outcome Measures were identified as secondary analysis in the study protocol, but are included to maintain consistency with other postings for this program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.